CLINICAL TRIAL: NCT00018395
Title: Cardiovascular Mortality Associated With Abnormal Calcium Metabolism
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: CADE-AI
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Disease; Kidney Disease
Keywords: Calcium Metabolism
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases

SUMMARY:
The purpose of this cohort study is to estimate the risk of cardiovascular mortality associated with abnormal calcium metabolism

ELIGIBILITY:
All ESRD patients who indicated dialysis in 1990-1993

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-08; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States